CLINICAL TRIAL: NCT03608241
Title: A PHASE 1, RANDOMIZED, OPEN LABEL, 2-WAY CROSSOVER STUDY TO ESTIMATE THE EFFECT OF MULTIPLE DOSE PF-06651600 ON THE PHARMACOKINETICS OF SINGLE DOSE ORAL CONTRACEPTIVE STEROIDS IN HEALTHY FEMALE SUBJECTS
Brief Title: A STUDY TO ESTIMATE THE EFFECT OF PF-06651600 ON THE PHARMACOKINETICS (PK) OF ORAL CONTRACEPTIVE (OC)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: B7981018
Record Dates: First submitted 2018-07-06; First posted 2018-07-31 (Actual); Last update posted 2019-04-09 (Actual); Status verified 2019-04

CONDITIONS: Healthy Females
Keywords: female; post-menopausal; healthy; oral contraceptive
MeSH Terms: interventions — PF-06651600; Ethinyl Estradiol; Contraceptives, Oral

STUDY DESIGN:
Masking Description: Open label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment sequence 1 (Experimental): Treatment sequence 1 will receive a single dose of an oral contraceptive during the first period of the study (period 1) and then continue to the second period (Period 2) of the study where they will receive PF-06651600 every day for 11 days and a single dose of an oral contraceptive towards the end of the period.
  Interventions: Drug: PF-06651600; Drug: Ethinyl estradiol (EE) and levonogestrel (LN)
- Treatment Sequence 2 (Experimental): Treatment sequence 2 will receive PF-06651600 every day for 11 days during the first period of the study (period 1) and a single dose of an oral contraceptive towards the end of this period. After completion of Period 1, there will be a washout period of at least 10 days before starting the second period of the study (period 2). During period 2, a single dose of an oral contraceptive will be received.
  Interventions: Drug: PF-06651600; Drug: Ethinyl estradiol (EE) and levonogestrel (LN)

INTERVENTIONS:
Drug: PF-06651600 — 200 mg by mouth (PO) Once daily (QD) for 11 days
Drug: Ethinyl estradiol (EE) and levonogestrel (LN) — Single dose of Oral tablet containing 30 ug EE and 150 ug of LN
  Other Names: Oral contraceptive

SUMMARY:
This is a Phase 1, randomized, 2 way crossover, multiple dose, open label study of the effect of multiple dose PF-06651600 on single dose OC PK in healthy female subjects. Subjects will be randomized to 1 of 2 treatment sequences.

ELIGIBILITY:
Inclusion Criteria

Subjects must meet all of the following inclusion criteria to be eligible for enrollment in the study:

1. Healthy female subjects of non childbearing potential

   Female subjects of non childbearing potential must meet at least 1 of the following criteria:
   1. Achieved postmenopausal status, defined as follows: cessation of regular menses for at least 12 consecutive months with no alternative pathological or physiological cause; and have a serum follicle stimulating hormone (FSH) level confirming the postmenopausal state;
   2. Have undergone a documented hysterectomy and/or bilateral oophorectomy;
   3. Have medically confirmed ovarian failure. All other female subjects (including female subjects with tubal ligations) are considered to be of childbearing potential and are not eligible for this study.
2. Body mass index (BMI) of 17.5 to 35 kg/m2; and a total body weight >50 kg (110 lb).

Exclusion Criteria

Subjects with any of the following characteristics/conditions will not be included in the study:

1. Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurological, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing).
2. History of drug abuse with less than 6 months of abstinence prior to the baseline visit.
3. History of regular alcohol consumption exceeding 7 drinks/week for female subjects (1 drink = 5 ounces [150 mL] of wine or 12 ounces [360 mL] of beer or 1.5 ounces [45 mL] of hard liquor) within 6 months before screening.
4. Any medical reason which would contraindicate the administration of oral contraceptives (as per the label) or history of discontinued use of oral contraceptives due to medical reasons.
5. Subjects with a known immunodeficiency disorder or a first degree relative with a hereditary immunodeficiency.
6. Subjects who have a malignancy or a history of malignancy, with the exception of adequately treated or excised non metastatic basal cell or squamous cell cancer of the skin or cervical carcinoma in situ.
7. Any current evidence of untreated active or latent or inadequately treated infection with Mycobacterium tuberculosis (TB).
8. History of human immunodeficiency virus (HIV), hepatitis B, or hepatitis C; positive testing

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Healthy female subjects of non childbearing potential
Enrollment: 12 (Actual)
Dates: Start 2018-09-21 (Actual); Primary Completion 2018-11-23 (Actual); Study Completion 2018-11-23 (Actual)

PRIMARY OUTCOMES:
Area Under the Curve From Time Zero to Extrapolated Infinite Time (AUCinf) for EE | 0 (pre-dose),1, 1.5. 2,4,6,8,12,24 and 48 hours post-dose
  AUCinf = Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0-inf). It is obtained from AUC (0-t) plus AUC (t-inf).
Area Under the Curve From Time Zero to Extrapolated Infinite Time (AUCinf) for LN | 0 (pre-dose), 1, 1.5, 2, 4, 6, 8, 12, 24 and 48 hours post-dose
  AUCinf = Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0-inf). It is obtained from AUC (0-t) plus AUC (t-inf).

SECONDARY OUTCOMES:
Number of Participants With Treatment Emergent Treatment-Related Adverse Events (AEs) | Baseline (Day 0) up to 28 days after last dose of study drug
Number of Adverse Events by Severity | Baseline up to 28 days after last dose
Number of Participants With Categorical Vital Signs Data | Baseline through study completion, approximately 23 days.
Number of Participants With Change From Baseline in Laboratory Tests Results | Baseline through study completion, approximately 23 days.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (2):
- United States (2):
  - Quotient Sciences, Coral Gables, Florida
  - Quotient Sciences-Miami, Inc., Miami, Florida

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B7981018&StudyName=A+Phase+1%2C+Randomized%2C+Open+Label%2C+2-way+Crossover+Study+To+Estimate+The+Effect+Of+Multiple+Dose+Pf-06651600+On+The+Pharmacokinetics+Of+Single+Dose+Oral+Contraceptive+Steroids+In+Healthy+Female+Subjects